CLINICAL TRIAL: NCT05541198
Title: Evaluation of Pressure Injury Prevention Care Bundle Application in Intensive Care Unit Patients Diagnosed With Internal Diseases
Brief Title: Prevention to Pressure Injury With Care Bundle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GALTAS
Record Dates: First submitted 2022-08-25; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-07

CONDITIONS: Pressure Injury
Keywords: Bundle care; Pressure injury; Intensive care; Nursing
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Routine clinical care continued to be provided to the patients in the control group.
  Routine maintenance applications include the following parameters;
  1. Risk assessment using Braden Risk Scale
  2. Positioning
  3. Elevate the heels.
- Intervention Group (Experimental): A pressure injury care bundle was developed in line with the relevant literature. After the development of the bundle, a 30-minute training program was applied to the nurses on general information about pressure injuries, the pressure injury care bundle, and how to use the bundle. The training program was carried out in four separate sessions arranged according to the working schedules of 40 nurses providing services in ICU.
  Care Bundle include this parameters;
  1. Risk Assessment
  2. Skin Assessment
  3. Skin Care
  4. Positioning
  5. Regulation of Nutrition and Liquid Management
  Interventions: Other: Pressure Injury Prevention Care Bundle

INTERVENTIONS:
Other: Pressure Injury Prevention Care Bundle — 1. Risk Assessment
  2. Skin Assessment
  3. Skin Care
  4. Positioning
  5. Regulation of Nutrition and Liquid Management
  Arms: Intervention Group

SUMMARY:
Aim: The study was conducted in order to evaluate of pressure injury prevention care bundle application in intensive care unit patients diagnosed with internal diseases.

Background: Although a pressure injury is a problem that requires treatment for a long time and takes time to heal, it is possible to prevent it with appropriate interventions. Evidence for the prevention of pressure injuries suggests using evidence-based guidelines or care bundles.

Design: Quasi-experimental and control group study. Methods: The study was conducted on 98 patients, 49 in the control group and 49 in the intervention group, diagnosed with internal diseases and hospitalized in the intensive care unit of a training and research hospital between July-December 2021. In the collection of the study data, patient information form, pressure injury prevention care bundle tool, and Braden Risk Scale were used. While routine clinical care continued to be provided to the patients in the control group, pressure injury prevention care bundle was applied to the patients in the intervention group.

DETAILED DESCRIPTION:
As preventing the development of pressure injury is a parameter that shows the quality of care, the most significant responsibility in preventing pressure injury belongs to nurses. Pressure injury develops as a result of inadequate nursing care and not routinely applying evidence-based planned care in preventing pressure injury. In this sense, nurses can prevent the development of pressure injury by evaluating the patient holistically and applying evidence-based preventive pressure injury care.

Although a pressure injury is a problem that requires treatment for a long time and takes time to heal, it is possible to prevent it with appropriate interventions.In this context, European Pressure Injury Advisory Panel (EPIAP) and National Pressure Injury Advisory Panel (NPIAP) determined several preventive stages in order to prevent pressure injuries, such as risk assessment, skin assessment and care, repositioning, using pressure reducing surfaces, protection from incontinence, nutrition and fluid support, and training .

Evidence for the prevention of pressure injuries suggests using evidence-based guidelines or care bundles. Care bundle is an organized and medical regulations-based set of applications that promotes compliance with guidelines and increases the quality of care by facilitating the provision of evidence-based care.

In the present study, it was aimed to prevent the development of pressure injuries by applying the prepared pressure injury prevention bundle care to the patients hospitalized in the intensive care unit patients diagnosed with internal diseases and thus to determine the effectiveness of the care bundle.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above,
* Who did not have any pressure injuries on any part of their body,
* Who were expected to stay in the clinic for at least 24 hours,
* Who were diagnosed with an internal disease

Exclusion Criteria:

* Who were younger than 18 years,
* Who had a pressure injury on any part of their body,
* Who were expected to stay in the clinic for less than 24 hours
* Who had intensive care indications other than an internal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | 60 minutes
  The form prepared by the researcher includes questions inquiring about the sociodemographic and background information of the patients, clinical characteristics and laboratory results.
Pressure Injury Prevention Care Bundle | 3-4 weeks
  Care bundle includes risk assessment, skin assessment, skin care, repositioning, regulating nutrition and fluid intake.
Braden Risk Assessment Tool | 1 hour
  With this tool, six parameters of the patient's stimulant perception, activity, mobility, the effect caused on the skin by humidity, friction, and shearing tension are measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Gülnaz Altaş, Istanbul, Istanbul, Uskudar, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: guidelines — https://www.epuap.org/pu-guidelines/
- See also: article — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5098472/
- See also: article — https://dergipark.org.tr/tr/pub/aktd/issue/28690/306004
- See also: article — http://www.yoihd.org.tr/sayfa.aspx?id=142.
- See also: article — https://dergipark.org.tr/en/pub/ausbid/issue/67542/1003094
- See also: article — https://dergipark.org.tr/en/pub/ataunihem/issue/2666/34584
- See also: article — https://pubmed.ncbi.nlm.nih.gov/24565372/
- See also: article — https://search.trdizin.gov.tr/yayin/detay/335810/
- See also: article — https://www.turkiyeklinikleri.com/article/tr-dekubit-ve-basi-ulserleri-85382.html
- See also: article — https://atif.sobiad.com/index.jsp?modul=makale-detay&Alan=saglik&Id=AWfsBFORHDbCZb_mQ-td

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT05541198/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT05541198/ICF_001.pdf